CLINICAL TRIAL: NCT00804544
Title: Tc-99m Sestamibi SPECT/CT for Prediction of the Response of Locally Advanced Breast Malignancy to Neoadjuvant Chemotherapy
Brief Title: 99mTc-MIBI SPECT/CT in Breast Malignancy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 4 patients have been enrolled into the pilot study. No complications reported. Another clinical trial has been designed.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Irina Rachinsky, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-08-383; 12967 (Other: REB)
Record Dates: First submitted 2008-12-04; First posted 2008-12-09 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: Integrated SPECT/CT; 99mTc-sestMIBI; Chemosensitivity
MeSH Terms: conditions — Breast Neoplasms | interventions — Single Photon Emission Computed Tomography Computed Tomography; Multimodal Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Mammoscintigraphy with SPECT-CT optimized 99mTc-MIBI imaging (experimental arm) will be compared to conventional planar imaging. Mammoscintigraphy results before and after chemotherapy and radiation therapy, will be compared to the histopathological results after surgery.
  Interventions: Device: SPECT/CT

INTERVENTIONS:
Device: SPECT/CT — SPECT/Low-Dose MultiSclice CT
  Other Names: Integrated SPECT/CT; Hybrid imaging

SUMMARY:
99mTc-SestaMIBI mammoscintigraphy (MMS) may be used in patients with locally advanced breast cancer (LABC) scheduled for neoadjuvant chemotherapy. MMS may be performed for 1) nodal staging of axillary lymph node metastases, 2) prediction of chemosensitivity or Pgp/MDR-1 mediated chemoresistance, and 3) evaluation of efficacy to chemotherapy and radiation therapy.

MMS is routinely performed with planar/SPECT imaging according to the Society of Nuclear Medicine and European Association of Nuclear Medicine guidelines.

In this pilot study, an optimised acquisition protocol will be setup with SPECT/low-dose multislice CT in addition to planar imaging.

DETAILED DESCRIPTION:
99mTc-SestaMIBI is a lipophylic cation as many cytotoxic chemotherapy drugs (i.e. anthracyclines, inhibitor of topoisomerase II, antimicrotubule, vinca alkaloids, inhibitors of DNA replication) accumulating in the mitochondria of tumour cells. MIBI tumour uptake is related to viability and proliferation due to increased perfusion and increased energy-dependent metabolism.

99mTc-SestaMIBI is a substrate for the glycoprotein P (Pgp) pump encoded by the multidrug resistance gene -1 (MDR-1). MIBI tumour uptake with no significant wash-out over time (<45% at 3H) predicts a chemosensitivity with no Pgp/MDR-1 overexpression. MIBI efflux with no significant tumour uptake predicts efflux of chemotherapy drugs from the tumour cells related to Pgp/MDR-1 overexpression or to anti-apoptotic Bcl-2 overexpression. Early MIBI efflux (< 1H) may also be related to pro-apoptotic Bax overexpression.

SPECT/CT will be used for anatomic localisation and and attenuation correction. CT from SPECT/CT is a low-dose (< 2 mSv) multislice CT (4 slice). SPECT/CT will also be used for correction of image-degrading factors including collimator-detector-response compensation for resolution recovery, and scatter correction. SPECT/CT based absolute semi-quantification of MIBI uptake into primary tumour and lymph nodes (i.e. standardised uptake value or SUV) will also be performed.

SPECT/CT optimised imaging will be compared to planar/SPECT conventional nuclear imaging for 1) detection of MIBI-avid primary breast tumour and lymph node metastases, 2) semi-quantification of MIBI uptake (T/B, SUV, and %wash-out) into primary breast tumour and lymph node metastases, 3) prediction of chemosensitivity at baseline, 3) Evaluation of chemotherapy efficacy after the first course of chemotherapy (after 2 weeks) compared to clinical response and histo-pathological response.

SPECT/CT mammoscintigraphy findings will be compared to clinical findings (palpation), radiological findings (mammography, US, MRI), and histo-pathological findings (Pgp/MDR-1 expression) into tumours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven breast cancer
* Patients with locally advanced breast cancer (stages T2-4 N0-3 M0)
* Patients scheduled for neoadjuvant chemotherapy
* Patients scheduled for radical modified mastectomy
* Patients with no physical and/or psychological contraindications
* Patients with no recent nuclear medicine study using long-lived isotopes (i.e. 67Ga, 111In, 131I) within the 48 hour preceding the mammoscintigraphy

Exclusion Criteria:

* Patient with no histologically proven breast cancer
* Patients with early stage T1 breast cancer
* Patients who are not candidates for neoadjuvant chemotherapy
* Patients who are not surgical candidates
* Patients with physical and/or psychological contraindications
* Pregnant or breast feeding patients
* Patients with a recent nuclear medicine study using long-lived isotopes (i.e. 67Ga, 111In, 131I) within the 48 hour preceding the mammoscintigraphy

Ages: 25 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
1- Nodal staging 2- Prediction of chemosensitivity 3- Evaluation of chemosensitivity | 1 year

SECONDARY OUTCOMES:
Added-Value of integrated SPECT/Low-dose MultiSlice CT versus planar/SPECT imaging in mammoscintigraphy with 99mTc-SestaMIBI | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Irina Rachinsky, MD, MSc, Principal Investigator — The UWO - LHSC - Department of Nuclear Medicine; Albert A Driedger, MD, PhD, Study Chair — The UWO -LHSC - Department of Nuclear Medicine; Muriel Brackstone, MD, Study Director — The UWO - LHSC - Department of General Surgery; Francisco Perera, MD, Study Director — The UWO - LHSC - Department of Medical Oncology
Locations (1):
- South Street Hospital - Department of Nuclear Medicine, London, Ontario, Canada

REFERENCES:
- [Background] Moretti JL, Hauet N, Caglar M, Rebillard O, Burak Z. To use MIBI or not to use MIBI? That is the question when assessing tumour cells. Eur J Nucl Med Mol Imaging. 2005 Jul;32(7):836-42. doi: 10.1007/s00259-005-1840-x. PMID 15902437
- [Background] Spanu A, Chessa F, Sanna D, Cottu P, Manca A, Nuvoli S, Madeddu G. Scintimammography with a high resolution dedicated breast camera in comparison with SPECT/CT in primary breast cancer detection. Q J Nucl Med Mol Imaging. 2009 Jun;53(3):271-80. Epub 2008 Jul 4. PMID 18596669
- [Background] Maini CL, Tofani A, Sciuto R, Semprebene A, Cavaliere R, Mottolese M, Benevolo M, Ferranti F, Grandinetti ML, Vici P, Lopez M, Botti C. Technetium-99m-MIBI scintigraphy in the assessment of neoadjuvant chemotherapy in breast carcinoma. J Nucl Med. 1997 Oct;38(10):1546-51. PMID 9379190
- [Background] Takamura Y, Miyoshi Y, Taguchi T, Noguchi S. Prediction of chemotherapeutic response by Technetium 99m--MIBI scintigraphy in breast carcinoma patients. Cancer. 2001 Jul 15;92(2):232-9. doi: 10.1002/1097-0142(20010715)92:23.0.co;2-g. PMID 11466674
- [Background] Del Vecchio S, Zannetti A, Ciarmiello A, Aloj L, Caraco C, Fonti R, Botti G, D'Aiuto G, Salvatore M. Dynamic coupling of 99mTc-MIBI efflux and apoptotic pathway activation in untreated breast cancer patients. Eur J Nucl Med Mol Imaging. 2002 Jun;29(6):809-14. doi: 10.1007/s00259-002-0773-x. Epub 2002 Mar 13. PMID 12029556
- [Background] Sciuto R, Pasqualoni R, Bergomi S, Petrilli G, Vici P, Belli F, Botti C, Mottolese M, Maini CL. Prognostic value of (99m)Tc-sestamibi washout in predicting response of locally advanced breast cancer to neoadjuvant chemotherapy. J Nucl Med. 2002 Jun;43(6):745-51. PMID 12050317
- [Background] Khalkhali I, Diggles LE, Taillefer R, Vandestreek PR, Peller PJ, Abdel-Nabi HH. Procedure guideline for breast scintigraphy. Society of Nuclear Medicine. J Nucl Med. 1999 Jul;40(7):1233-5. No abstract available. PMID 10405150
- [Background] Xu HB, Li L, Xu Q. Tc-99m sestamibi scintimammography for the diagnosis of breast cancer: meta-analysis and meta-regression. Nucl Med Commun. 2011 Nov;32(11):980-8. doi: 10.1097/MNM.0b013e32834b43a9. PMID 21956488
- [Background] Schillaci O, Danieli R, Filippi L, Romano P, Cossu E, Manni C, Simonetti G. Scintimammography with a hybrid SPECT/CT imaging system. Anticancer Res. 2007 Jan-Feb;27(1B):557-62. PMID 17348441
- [Background] Goldsmith SJ, Parsons W, Guiberteau MJ, Stern LH, Lanzkowsky L, Weigert J, Heston TF, Jones E, Buscombe J, Stabin MG; Society of Nuclear Medicine. SNM practice guideline for breast scintigraphy with breast-specific gamma-cameras 1.0. J Nucl Med Technol. 2010 Dec;38(4):219-24. doi: 10.2967/jnmt.110.082271. Epub 2010 Nov 5. No abstract available. PMID 21057112
- [Result] Bombardieri E, Aktolun C, Baum RP, Bishof-Delaloye A, Buscombe J, Chatal JF, Maffioli L, Moncayo R, Mortelmans L, Reske SN. Breast scintigraphy: procedure guidelines for tumour imaging. Eur J Nucl Med Mol Imaging. 2003 Dec;30(12):BP107-14. doi: 10.1007/s00259-003-1354-3. No abstract available. PMID 14989223
- See also: The University of Western Ontario — http://www.uwo.ca/